CLINICAL TRIAL: NCT03279588
Title: Diagnostic Accuracy and Role of Bedside Ultrasound in Patients With Suspected Acute Diverticulitis
Brief Title: Diagnostic Accuracy of Bedside Ultrasound in Suspected Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 11004
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Diverticulitis; Abdominal Pain
Keywords: Ultrasound diagnosis; Abdominal Ultrasound; Emergency Department
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bedside Ultrasound — Patients presenting to the Emergency Department with abdominal pain suspected of acute diverticulitis are evaluated with standard care by an Emergency Physician (tutor); at the time the tutor requests an imaging test performed by Radiologist (CT scan or US scan), he notifies another physicians skilled in bedside abdominal US (ultrasonographer), who evaluates the patient and performs the US scan. Ultrasonographer after completation of US and knowing blood samples results fills in a standardized form reporting the diagnostic hypotesis, the need for additional work-up (if deemed necessary), and the disposition of the patient. The standardized form completed by the ultrasonographer will be compared with the actual management of the patient.

SUMMARY:
Colonic diverticulitis is a common clinical condition in patients presenting to the Emergency Department (ED) with abdominal pain. The diagnosis and staging of patients with suspected acute diverticulitis is often made by CT imaging with intravenous contrast, which involves radiation exposure, is expensive and has contraindications. The aim of this study is to evaluate the diagnostic accuracy and role of bedside abdominal US for the diagnosis of acute diverticulitis

DETAILED DESCRIPTION:
Colonic diverticulitis is a common clinical condition; about 20% of patients with colonic diverticulosis experience abdominal symptoms and, eventually, complications such as episodes of diverticulitis or bleeding. The distinction between patients with uncomplicated or complicated diverticulitis affects the clinical management: medical therapy for the first, interventional therapy for the latter. CT imaging with intravenous contrast has become the gold standard in the diagnosis and staging of patients with suspected acute diverticulitis but, unfortunately, CT involves radiation exposure, is expensive and has contraindications. UltraSound (US) is a real-time dynamic examination with wide availability and easy accessibility and may be useful in diagnosing and managing critically ill patients who cannot be moved to CT. In a recent meta-analysis, US exam performed by Radiologists showed a pooled sensitivity of 90% (vs 95% for CT, p = 0.86) and a specificity of 90% (vs 96% for CT, p = 0.04). US is increasingly used at bedside to rapidly assess patients presenting to the Emergency Department. No previous studies have investigated the diagnostic accuracy of abdominal US performed by physician at bedside as an extension of physical examination. This study evaluates the diagnostic accuracy of bedside abdominal US.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained
* patients with abdominal pain presenting to the Emergency Department with a suspicon of diverticular disease, in whom the tutor physician orders an imaging study (abdominal CT or abdominal US performed by the Radiologist)

Exclusion Criteria:

* no ultrasonographer physician who can perform bedside abdominal US is present
* the patient does not undergo imaging study
* clinical conditions of the patient are particularly severe, preventing an adequate enrollment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every patient presenting with symptoms suspected of diverticular disease to the Emergency Department of four Italian hospitals will be considered eligible for the study
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of bedside abdominal US performed by Emergency Physicians for the diagnosis and stratification of acute diverticulitis | 30 days
  Sensitivity, specificity, negative and positive predictive value, negative and positive likelihood ratio of bedside abdominal US performed by Emergency Physicians for the diagnosis of acute diverticulitis.

SECONDARY OUTCOMES:
Management of patient | 30 days
  To evaluate the reliability of the management proposed by the ultrasonographer on the basis of clinical, laboratoristic and ultrasonographic data.
Time reduction | 30 days
  To evaluate if the use of bedside abdominal US performed by Emergency Physicians can reduce the time needed for the diagnosis
CT scan reduction | 30 days
  To evaluate if the use of bedside abdominal US performed by Emergency Physicians can raduce the number of CT scans performed in patients with suspected acute diverticulitis

CONTACTS AND LOCATIONS:
Overall Officials: Peiman Nazerian, MD, Principal Investigator — Emergency Departmet Azienda Ospedaliero Universitaria Careggi
Locations (4):
- Italy (4):
  - Department of Emergency Medicine, Figline Valdarno, Firenze
  - Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Emergency Department ASST degli Spedali Civili di Brescia, Brescia
  - Emergency Department Nuovo Ospedale di Prato, Prato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sartelli M, Catena F, Ansaloni L, Coccolini F, Griffiths EA, Abu-Zidan FM, Di Saverio S, Ulrych J, Kluger Y, Ben-Ishay O, Moore FA, Ivatury RR, Coimbra R, Peitzman AB, Leppaniemi A, Fraga GP, Maier RV, Chiara O, Kashuk J, Sakakushev B, Weber DG, Latifi R, Biffl W, Bala M, Karamarkovic A, Inaba K, Ordonez CA, Hecker A, Augustin G, Demetrashvili Z, Melo RB, Marwah S, Zachariah SK, Shelat VG, McFarlane M, Rems M, Gomes CA, Faro MP, Junior GA, Negoi I, Cui Y, Sato N, Vereczkei A, Bellanova G, Birindelli A, Di Carlo I, Kok KY, Gachabayov M, Gkiokas G, Bouliaris K, Colak E, Isik A, Rios-Cruz D, Soto R, Moore EE. WSES Guidelines for the management of acute left sided colonic diverticulitis in the emergency setting. World J Emerg Surg. 2016 Jul 29;11:37. doi: 10.1186/s13017-016-0095-0. eCollection 2016. PMID 27478494
- [Background] Cuomo R, Barbara G, Pace F, Annese V, Bassotti G, Binda GA, Casetti T, Colecchia A, Festi D, Fiocca R, Laghi A, Maconi G, Nascimbeni R, Scarpignato C, Villanacci V, Annibale B. Italian consensus conference for colonic diverticulosis and diverticular disease. United European Gastroenterol J. 2014 Oct;2(5):413-42. doi: 10.1177/2050640614547068. PMID 25360320
- [Background] Andeweg CS, Wegdam JA, Groenewoud J, van der Wilt GJ, van Goor H, Bleichrodt RP. Toward an evidence-based step-up approach in diagnosing diverticulitis. Scand J Gastroenterol. 2014 Jul;49(7):775-84. doi: 10.3109/00365521.2014.908475. Epub 2014 May 30. PMID 24874087
- [Background] Lameris W, van Randen A, Bipat S, Bossuyt PM, Boermeester MA, Stoker J. Graded compression ultrasonography and computed tomography in acute colonic diverticulitis: meta-analysis of test accuracy. Eur Radiol. 2008 Nov;18(11):2498-511. doi: 10.1007/s00330-008-1018-6. Epub 2008 Jun 4. PMID 18523784
- [Background] Liljegren G, Chabok A, Wickbom M, Smedh K, Nilsson K. Acute colonic diverticulitis: a systematic review of diagnostic accuracy. Colorectal Dis. 2007 Jul;9(6):480-8. doi: 10.1111/j.1463-1318.2007.01238.x. PMID 17573739
- [Background] Mazzei MA, Cioffi Squitieri N, Guerrini S, Stabile Ianora AA, Cagini L, Macarini L, Giganti M, Volterrani L. Sigmoid diverticulitis: US findings. Crit Ultrasound J. 2013 Jul 15;5 Suppl 1(Suppl 1):S5. doi: 10.1186/2036-7902-5-S1-S5. Epub 2013 Jul 15. PMID 23902791